CLINICAL TRIAL: NCT04213378
Title: Evaluation of the Efficacy and Safety of a Paclitaxel Eluting PTCA Balloon Catheter in Coronary In-stent Restenosis: a Randomized, Open-label, Positive Parallel Controlled, Multicenter Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of a Paclitaxel Eluting PTCA Balloon Catheter in Coronary In-stent Restenosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: West China Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); The Third Xiangya Hospital of Central South University (Other); Hebei Medical University Third Hospital (Other); TEDA International Cardiovascular Hospital (Other); Tianjin People's Hospital (Other); The Second Hospital of Shandong University (Other); Hainan People's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Shanghai Chest Hospital (Other); Renmin Hospital of Wuhan University (Other); Taizhou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU CT016
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Coronary In-stent Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Paclitaxel eluting PTCA balloon (Experimental): Treatment of coronary in-stent restenosis with paclitaxel eluting PTCA balloon
  Interventions: Device: Paclitaxel eluting PTCA balloon
- SeQuent® Please paclitaxel eluting balloon (Active Comparator): Treatment of coronary in-stent restenosis with SeQuent® Please paclitaxel eluting balloon
  Interventions: Device: SeQuent® Please paclitaxel eluting balloon

INTERVENTIONS:
Device: Paclitaxel eluting PTCA balloon — Treatment of coronary in-stent re-stenosis with paclitaxel eluting PTCA balloon
  Arms: Paclitaxel eluting PTCA balloon
Device: SeQuent® Please paclitaxel eluting balloon — Treatment of coronary in-stent re-stenosis with SeQuent® Please paclitaxel eluting balloon
  Arms: SeQuent® Please paclitaxel eluting balloon

SUMMARY:
Over the past two decades, stents implantation has developed as a standard treatment for coronary stenosis lesions. However, int-stent restenosis (ISR) was one of the main factors affecting the long-term efficacy of coronary artery interventional therapy, with the incidence of ISR after percutaneous coronary intervention ranging from 5% to 35%. At present, there are three main means for ISR: (1) simple balloon dilation; 2) intravascular radiotherapy; and (3) drug elution stent. But the results are still not ideal. Drug coated balloon (DCB) is a new method that may be used to treat ISR in recent years. In the PEPCAD II study, when dealing with ISR, the paclitaxel eluting balloon (PEB) SeQuent® Please significantly reduced the major adverse cardiovascular events (MACEs) compared to the paclitaxel eluting stent (PES) TAXUS Liberte. In ISR-I and ISR-II trial, it was found that compared with uncoated PTCA balloons, PEB could significantly inhibit endothelial hyperplasia and significantly reduce MACEs treating ISR. The purpose of this study was to assess the efficacy and safety of a Chinese-developed PEB in treatment of coronary ISR compared to SeQuent® Please PEB.

ELIGIBILITY:
Inclusion Criteria:

* Patients oriented

  1. Patients with age between 18 and 80 years old (including 18 and 80 years old);
  2. Patients with stable angina, or unstable angina pectoris, or old myocardial infarction (MI) or with evidence of local myocardial ischemia although without symptoms;
  3. Patients with restenosis after the first time stent implantation of de novo coronary lesions (i.e., no other surgical treatments for the target lesions except for the first stent implantation);
  4. Patients with the willing to receive their own coronary angioplasty;
  5. Patients with LVEF>30% measured within 30 days before recruitment;
  6. Patients agree to receive 9-month angiography follow-up, and agree to receive 30 days, 6 months, 12 months clinical follow-up;
  7. Patients at the age of childbirth must take effective contraception measures until the study is completed since they are chosen into screening period;
  8. Patients agree to take part in the trial and sign the informed consent.
* Lesions oriented (Visual estimation)

  1. Patients with Mehran type I, type II and type III in-stent restenosis (ISR);
  2. Reference vascular diameter between 2.0-4.0 mm (including 2.0 and 4.0 mm), length<30mm;
  3. The percent of lumen ISR ≥70%, or ≥50% with local ischemia evidence before interventional surgery;
  4. Patients with residual stenosis ≤30%, and ≤ type B dissection post pretreatment;
  5. Distance between other lesions that require treatment and target lesions >10 mm;
  6. Patients with coronary artery anatomy allowing delivery of research device to target lesions.

Exclusion Criteria:

* Patients oriented

  1. Subjects with consistent clinical symptoms and/or ECG changes and/or cardiac enzymes changes with MI (including STEMI and Non-STEMI) within one week;
  2. Subjects with cardiac shock, hemodynamic instability or refractory ventricular arrhythmia that require positive inotropic drugs or mechanical circulation support;
  3. Subjects with one of following conditions (from screening period to the day of operation): (1) life expectancy is less than 1 year because of other severe diseases (like cancer), (2) drug abuse at present (like alcohol, cocaine, heroin and so on), (3) plan to accept surgery that may cause the programs not to be complied with or confusing with data understanding;
  4. Subjects with bleeding diathesis or active gastrointestinal ulcers, or stroke/transient ischemic attack within 3 months;
  5. Subjects with severe congestive heart failure or severe heart failure at the level of NYHA IV;
  6. Subjects are receiving dialysis or baseline serum creatinine levels>2.0 mg/dL(177μmol/L);
  7. Subjects with severe valvular heart disease;
  8. Subjects who have been or are scheduled for a heart transplantation during the trial;
  9. Subjects who have been pregnant or is planning to be pregnant or is breastfeeding during the trial;
  10. Subjects who are participating in any other clinical trial;
  11. Researchers don't think they're suitable for the trial because of other reasons;
* Lesions oriented (Visual estimation)

  1. Total occlusion with TIMI 0 (Mehran IV stenosis);
  2. With the evidence of widespread thrombi in the target vessels prior to intervention;
  3. Planning to treat >3 lesions (i.e., up to 3 target lesions);
  4. Planning to treat >2 major epicardial vessels (i.e., up to 2 target lesions);
  5. Planning to treat a single lesions with more than 1 balloon;
  6. Planning to treat a true bifurcation lesion with double stents technique;
  7. Left main lesions.
* Combined medication oriented

  1. Subjects known to intolerant to dual antiplatelet therapy for 3 months post interventional treatment (e.g., aspirin and/or ticagrelor and/or clopidogrel);
  2. Subjects with leukopenia (WBC<3x10^9/L for more than 3 days) or neutropenia (NEUT<1x10^9/L for more than 3 days) or a history of platelet reduction (PLT 30x10^9/L);
  3. Subjects known to be intolerant or allergic to paclitaxel.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of target lesion late lumen loss | 9 months

SECONDARY OUTCOMES:
Rate of interventional therapy success | 0-24 hours, 30 days, 6 months, 9 months, 12 months
  Including rate of device success, rate of disease success and rate of clinical success
Rate of target lesion restenosis | 9 months
Device-oriented composite clinical cardiovascular outcomes | 30 days, 6 months, 9 months, 12 months
  Cardiac death, target vessel-related myocardial infarction, symptoms-driven target lesion revascularization
Patient-oriented composite clinical cardiovascular outcomes | 30 days, 6 months, 9 months, 12 months
  All-cause mortality, all myocardial infarction, all revascularization
Rate of ARC defined thrombosis events | 0-24 hours, 30 days, 6 months, 9 months, 12 months
  All definite, probable and possible thrombosis in acute, subacute and late stage

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD, PhD, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Xue W, Ma J, Yu X, Ruan Z, Sun Y, Wu T, Zhang X, Wu L. Analysis of the incidence and influencing factors associated with binary restenosis of target lesions after drug-coated balloon angioplasty for patients with in-stent restenosis. BMC Cardiovasc Disord. 2022 Nov 20;22(1):493. doi: 10.1186/s12872-022-02923-z. PMID 36404303